CLINICAL TRIAL: NCT04388904
Title: A Phase 4, Single-arm, Open-label Study to Evaluate the Efficacy and Safety of Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (D/C/F/TAF) Once Daily Fixed-dose Combination (FDC) Regimen in Antiretroviral Treatment-experienced Human Immunodeficiency Virus Type 1 (HIV-1) Infected Subjects Not Currently Receiving Any Antiretroviral Therapy.
Brief Title: Rapid Reinitiation of a Single Tablet Antiretroviral Therapy Using Symtuza® in HIV-1 Infected Treatment-Experienced Patients Off Therapy. (ReSTART)
Acronym: ReSTART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Crofoot Research Center, Inc. (Industry)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMC114FD2HTX4007
Record Dates: First submitted 2020-05-12; First posted 2020-05-14 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: HIV-1-infection
Keywords: Acquired Immunodeficiency Syndrome; HIV Infections; Sexually Transmitted Diseases, Viral; Anti-Retroviral Agents; Antiviral Agents
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Sexually Transmitted Diseases, Viral | interventions — Darunavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (FDC) (Experimental): Participants will receive oral tablet containing Darunavir 800 milligram (mg)/ Cobicistat 150 mg/ Emtricitabine 200 mg/ Tenofovir Alafenamide 10 mg (D/C/F/TAF) fixed-dose combination (FDC) once daily within 24 hours of the screening/baseline visit.
  Interventions: Drug: Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (FDC)

INTERVENTIONS:
Drug: Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (FDC) — Participants will receive Symtuza®. An oral tablet containing Darunavir 800 mg /Cobicistat 150 mg /Emtricitabine 200 mg /Tenofovir Alafenamide 10 mg FDC, once daily within 24 hours of the screening/ baseline visit.

SUMMARY:
The purpose of this study is to demonstrate the effectiveness of Symtuza® in a rapid reinitiation model of care in patients with HIV-1 infection and who are treatment-experienced but have been off of antiretroviral therapy (ART) for 12 or more weeks.

DETAILED DESCRIPTION:
In the United States, only 49 percent of persons living with HIV infection are currently retained in care (Centers for Disease Control, 2018). Many individuals initially start antiretroviral therapy (ART) but fall out of care and discontinue treatment, only to reenter care at a later date. Gaps in care contribute to the likelihood that a patient might not have a recent viral load or CD4 count, as well as knowledge of previous ART regimens or resistance data. Furthermore, high plasma HIV-1 RNA is a major risk factor for HIV transmission, and effective ART can reduce viremia and transmission of HIV to sexual partners by more than 96% (Cohen et al., 2011; Palella et al., 1998). Thus, a secondary goal of ART is to reduce the risk of HIV transmission.

Traditional models of care have an initial period where a person is brought back into care and assessed by a healthcare provider on various factors, including HIV RNA level, genotypic/ phenotypic resistance, immune status, renal/hepatic function, and general medical comorbidities before reinitiating ART. These steps can add weeks without treatment and, in turn, delay resupression of the virus and immune system improvement, as well as continuing to contribute to the community viral load and offering more opportunities for the person to fall out of care again. (Horburg et al., 2013) This traditional model places a burden on both the patient and the healthcare system as multiple visits are required, each one a potential point where the patient can be lost again to follow-up.

A rapid reinitiation of ART for persons who have fallen out of care is a potential intervention that could improve retention rates, patient satisfaction, and clinical outcomes. Given these factors, the single-tablet regimen of D/C/F/TAF (Symtuza®) may serve as an ideal regimen for a Rapid Reinitiation model of care, combining potency, sustained efficacy, a high genetic barrier to resistance, with a well-described safety profile of the individual components, and practical, convenient dosing.

This prospective, multicenter study will follow subjects for 48 weeks with subjects either returning to the site or having a virtual visit (TeleVisit) for Weeks 2, 4, 12, 24, 36, and 48. Baseline safety labs will dictate whether the ART regimen will need to be modified but will not be required to be completed at the initiation of ART. Assessment of drug accountability, reasons for non-adherence, recording of concomitant therapies, adverse events, weight, physical examinations (complete or symptom-directed), laboratory evaluations (for efficacy and safety), and health outcome assessments will be performed from baseline onwards.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at screening/baseline visit.
* Antiretroviral treatment-experienced and have not received any anti-HIV treatment within 12 weeks prior to screening.
* Contraceptive use by men or women should be consistent with the local regulations regarding the use of contraceptive methods for subject participating in clinical studies.
* Men must agree not to donate sperm during the study until 90 days after receiving the last dose of study drug (or longer, if dictated by local regulations).
* Must be able to swallow whole tablets or swallow tablets cut into halves.

Exclusion Criteria:

* Known active cryptococcal infection, active toxoplasmic encephalitis, Mycobacterium tuberculosis infection, or another AIDS-defining condition that in the judgment of the investigator would increase the risk of morbidity or mortality.
* Known resistance to any of the components of D/C/F/TAF; subjects with known or identified FTC resistance attributed to an M184V mutation alone will be permitted to remain in the study.
* Prior virologic failure on a DRV-containing regimen from known history or from medical records.
* Known history of clinically relevant hepatic disease or hepatitis that in the investigator's judgment is not compatible with D/C/F/TAF.
* Known history of severe hepatic impairment as diagnosed based on documented history of severe hepatic impairment (Child-Pugh C).
* Known history of chronic (≥3 months) renal insufficiency, defined as having an eGFR<30 mL/min according to the MDRD formula.
* Pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study or within 90 days after the last dose of study treatment.
* Plans to father a child while enrolled in this study or within 90 days after the last dose of study treatment.
* Current alcohol or substance use judged by the investigator to potentially interfere with subject study adherence.
* Known history of malignancy within the past 5 years or ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, noninvasive cutaneous squamous carcinoma.
* Known active, severe infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy that in the judgment of the investigator would increase the risk of morbidity or mortality.
* Any other condition or prior therapy for which, in the opinion of the investigator, participation would not be in the best interest of the subject (e.g., compromise the wellbeing) or that could prevent, limit, or confound the protocol-specified assessments.
* Subject unlikely to comply with the protocol requirements based on clinical judgment.
* Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 90 days before the planned first dose of study treatment or is currently enrolled in an investigational study.
* Subjects receiving ongoing therapy with contraindicated, not recommended, drugs that cannot be adequately dose-adjusted, or subjects with any known allergies to the excipients of the D/C/F/TAF.
* Employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of the employees or the investigator, or employees of Johnson & Johnson.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects who have HIV-1 RNA <50 copies/mL at week 48 | 48 week
  The proportion of subjects who have HIV-1 RNA <50 copies/mL at week 48 as defined by the FDA snapshot analysis (ITT)

SECONDARY OUTCOMES:
Proportion of subjects who have HIV-1 RNA <50 copies/mL at week 48 | Week 48
  Proportion of subjects who have HIV-1 RNA <200 copies/mL at week 48 as defined by the per-protocol (PP) analysis set
Proportion of subjects who have HIV-1 RNA <50 copies/mL at week 48 | Week 48
  Proportion of subjects who have HIV-1 RNA <200 copies/mL at week 48 as defined by the FDA snapshot analysis (ITT)
Proportion of subjects who have HIV-1 RNA <200 copies/mL at week 24 | Week 24
  Proportion of subjects who have HIV-1 RNA <200 copies/mL at week 24 as defined by the FDA snapshot analysis (ITT)
Change from baseline in HIV-1 RNA viral load | Weeks 24 and 48
  Change from baseline in log10 HIV-1 RNA viral load at Weeks 24 and 48
Change in baseline CD4 cell count | Weeks 12, 24, and 48
  Change in baseline CD4 cell count at Weeks 12, 24, and 48
Discontinuation after enrollment based on study stopping rules | Week 48
  Proportion of subjects that required discontinuation after enrollment based on study stopping rules
Discontinuation due to adverse events | Week 48
  Proportion of subjects discontinuing therapy due to adverse events
Proportion of subjects experiencing grade 3 and 4 adverse events | Week 48
  Proportion of subjects experiencing grade 3 and 4 adverse events
Proportion of subjects experiencing serious adverse events | Week 48
  Proportion of subjects experiencing serious adverse events
Proportion of subjects experiencing grade 3 and 4 laboratory abnormalities | Week 48
  Proportion of subjects experiencing grade 3 and 4 laboratory abnormalities
Proportion of subjects meeting resistance stopping rules requiring discontinuation of study drugs due baseline resistance findings | Week 48
  Proportion of subjects meeting resistance stopping rules requiring discontinuation of study drugs due baseline resistance findings
Proportion of subjects with baseline RT, INI, and PR (primary and secondary) RAMs | Week 48
  Proportion of subjects with baseline RT, INI, and PR (primary and secondary) RAMs
Proportion of subjects developing RAMs and loss of phenotypic susceptibility, when available, upon meeting PDVF | Week 48
  Proportion of subjects developing RAMs and loss of phenotypic susceptibility, when available, upon meeting PDVF
Proportion of subjects with PDVF at Week 24 and Week 48 | Weeks 24 and 48
  Proportion of subjects with PDVF at Week 24 and Week 48
Proportion of subjects lost to follow-up throughout the 48 Weeks of treatment | Week 48
  Proportion of subjects lost to follow-up throughout the 48 Weeks of treatment
Proportion of subjects taking study drug at Week 48 who have a documented clinic visit with a healthcare provider within 90 days of Week 48 visit. | Week 48
  Proportion of subjects taking study drug at Week 48 who have a documented clinic visit with a healthcare provider within 90 days of Week 48 visit.
Mean total satisfaction scores on the HIVTSQs at Weeks 4, 24, and 48 | Weeks 4, 24, and 48
  Mean total satisfaction scores on the HIVTSQs at Weeks 4, 24, and 48
Mean total depression scores on the PHQ-9 at baseline and Weeks 4, 24, and 48 | Weeks 4, 24, and 48
  Mean total depression scores on the PHQ-9 at baseline and Weeks 4, 24, and 48
Adherence as measured by pill count at Weeks 4, 12, 24, and 48 | Weeks 4, 12, 24, and 48
  Adherence as measured by pill count at Weeks 4, 12, 24, and 48

CONTACTS AND LOCATIONS:
Locations (1):
- The Crofoot Research Center, Inc., Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen MS, Chen YQ, McCauley M, Gamble T, Hosseinipour MC, Kumarasamy N, Hakim JG, Kumwenda J, Grinsztejn B, Pilotto JH, Godbole SV, Mehendale S, Chariyalertsak S, Santos BR, Mayer KH, Hoffman IF, Eshleman SH, Piwowar-Manning E, Wang L, Makhema J, Mills LA, de Bruyn G, Sanne I, Eron J, Gallant J, Havlir D, Swindells S, Ribaudo H, Elharrar V, Burns D, Taha TE, Nielsen-Saines K, Celentano D, Essex M, Fleming TR; HPTN 052 Study Team. Prevention of HIV-1 infection with early antiretroviral therapy. N Engl J Med. 2011 Aug 11;365(6):493-505. doi: 10.1056/NEJMoa1105243. Epub 2011 Jul 18. PMID 21767103
- [Background] Palella FJ Jr, Delaney KM, Moorman AC, Loveless MO, Fuhrer J, Satten GA, Aschman DJ, Holmberg SD. Declining morbidity and mortality among patients with advanced human immunodeficiency virus infection. HIV Outpatient Study Investigators. N Engl J Med. 1998 Mar 26;338(13):853-60. doi: 10.1056/NEJM199803263381301. PMID 9516219
- [Background] Centers for Disease Control and Prevention. Monitoring selected national HIV prevention and care objectives by using HIV surveillance data-United States and 6 dependent areas, 2016. HIV Surveillance Supplemental Report 2018;23(No. 4). http://www.cdc.gov/hiv/library/reports/ hiv-surveillance.html. Accessed [February 4, 2020]
- [Background] Horberg MA, Hurley LB, Silverberg MJ, Klein DB, Quesenberry CP, Mugavero MJ. Missed office visits and risk of mortality among HIV-infected subjects in a large healthcare system in the United States. AIDS Patient Care STDS. 2013 Aug;27(8):442-9. doi: 10.1089/apc.2013.0073. Epub 2013 Jul 19. PMID 23869466